CLINICAL TRIAL: NCT06953401
Title: Muscle Activity of the Gastrocnemius and Soleus Muscles During a Specific Contraction Task Assessed by Surface Electromyography
Brief Title: Muscle Activity of the Gastrocnemius and Soleus Muscles by Surface Electromyography.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Investigator, University of Extremadura
Other Study IDs: 150425
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Muscle Activity; Electromyography; Lower Limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Muscle contraction protocol for electromyographic assessment — Participants will perform a set of standardized lower limb muscle contractions (isometric, concentric, and eccentric) involving the gastrocnemius and soleus muscles while lying on an examination table and in standing position both static and dynamic as well as walking. Surface electromyography (mDurance® sEMG system) will be used to record muscle activation during each phase. The task is designed for physiological measurement only and does not constitute a therapeutic intervention. Protocol includes 3 trials per muscle and side, using standardized test conditions.

SUMMARY:
This cross-sectional, comparative study aims to evaluate and compare the surface electromyographic (sEMG) activity of the gastrocnemius (medial and lateral) and soleus muscles during static and dynamic contraction tasks. Participants will perform three tests-resting state, isometric, concentric, and eccentric contraction, and dynamic gait-with bilateral measurements. A subgroup analysis will examine muscle activity variations based on foot posture, using the Foot Posture Index (FPI). The study uses the validated mDurance® sEMG system to obtain objective data under controlled lab conditions. The findings will enhance understanding of the functional role of each muscle and could inform rehabilitation and injury prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years.
* No history of severe musculoskeletal disorders in the lower limbs.
* No recent surgery or injury in the last 6 months.
* No dermatological conditions affecting electrode placement.
* Not allergic to adhesives.
* Ability to perform the task without limitation.

  •. No high-intensity exercise in the 12 hours before testing
* Ability to provide informed consent and complete the assessment

Exclusion Criteria:

* Reduced lower limb mobility.
* Neuromuscular or skeletal conditions affecting the calf region.
* Intense physical activity 12 hours before testing.
* Lack of informed consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of healthy young adults enrolled in undergraduate programs at the Centro Universitario de Plasencia, University of Extremadura (Spain). Participants will be recruited through internal communication channels at the university. All participants will voluntarily agree to take part in the study and sign an informed consent form. Eligibility criteria include individuals aged 18 to 30 years, with no history of recent musculoskeletal injuries or surgeries in the lower limbs, and able to perform the required physical tasks without restriction. Subjects with foot postural alterations will also be included for later comparison with subjects without foot postural alterations.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle activation, microvolts (μV) | Baseline or Day 1. During a single assessment session (~30 minutes).
  Muscle activation (μV) as recorded by mDurance® sEMG system during the contraction protocol (soleus vs. gastrocnemius).

SECONDARY OUTCOMES:
RMS (root mean square) and peak EMG signal values (μV) | Baseline or Day 1. During the same assessment session
  RMS and peak EMG signal values (μV): average muscle activity measured by RMS (root mean square) and maximum voluntary contraction by peak activation. Comparison of Medial vs. Lateral Gastrocnemius Activation. Comparison of Medial vs. Lateral Gastrocnemius Activation
Differences in muscle activity by contraction type (μV) | Baseline or Day 1. Immediately after the execution of each contraction type during the session
  Differences in muscle activity by contraction type (μV): Effect of contraction type (isometric/concentric/eccentric) on muscle activity. Comparison of Medial vs. Lateral Gastrocnemius Activation
Activity differences by foot posture (pronated, neutral, supinated) | Baseline or Day 1. Immediately after foot posture assessment during the same session
  Muscle activation of the gastrocnemius and soleus will be compared based on foot posture (pronated, neutral, or supinated). This aims to identify whether foot type influences activation patterns.
Correlation with physical activity level Physical Activity Questionnaire (IPAQ-short version) | Baseline or Day 1. Collected at baseline before EMG assessment
  Correlation with physical activity level (IPAQ-short version): Correlation with sociodemographic and anthropometric factors (age, sex, BMI, activity level). Self-reported questionnaire assessing physical activity over the last 7 days. Physical activity is categorized as Low, Moderate, or High based on total MET-minutes/week. Sitting time is recorded separately as an indicator of sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: María Victoria CM María Victoria Cáceres Madrid, PhD, Principal Investigator — Departamento de Enfermería. Centro Universitario de Plasencia. Universidad de Extremadura; Olga LR Olga López Ripado, MSc, Principal Investigator — Departamento de Anatomía, Biología Celular y Zoología. Centro Universitario de Plasencia. Universidad de Extremadura; Alejando CP Alejandro Caña Pino, PhD, Principal Investigator — Departamento de Terapéutica Médico-Quirúrgica. Facultad de Enfermería y Terapia Ocupacional. Universidad de Extremadura; Marina FJ Fontán Jiménez, PhD, Principal Investigator — Departamento de Enfermería. Centro Universitario de Plasencia. Universidad de Extremadura; Raquel MA Raquel Mayordomo Acevedo, PhD, Study Director — Departamento de Anatomía, Biología Celular y Zoología. Centro Universitario de Plasencia. Universidad de Extremadura
Locations (1):
- Centro Universitario de Plasencia, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No